CLINICAL TRIAL: NCT04496414
Title: A Multi-center, Retrospective Registry Study on the Safety of Bactiseal Catheter
Brief Title: Bactiseal Catheter Safety Registry in China
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: C-BSEAL-001
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Results first posted 2021-12-21 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-02

CONDITIONS: Hydrocephalus
Keywords: hydrocephalus shunt; infection
MeSH Terms: conditions — Hydrocephalus; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Bactiseal Catheter — Bactiseal Catheter manufactured by Codman & Shurtleff, Inc. in the United States is a silicon catheter impregnated in rifampicin and clindamycin.

SUMMARY:
Research Purpose: This study aimed to continue to evaluate safety information from subjects implanted with a catheter (trade name: Bactiseal) produced by Codman & Shurtleff, Inc. of the United States. Device safety would be assessed based on all the adverse events that occurred within one year after the subjects implanted the catheter.

DETAILED DESCRIPTION:
This study aimed to continue to evaluate safety information from subjects implanted with a catheter (trade name: Bactiseal) produced by Codman & Shurtleff, Inc. of the United States. Device safety would be assessed based on all the adverse events that occurred within one year after the subjects implanted the catheter.

This study was designed to be single arm, multi-center, and retrospective. A total of 50 patients would be retrospectively enrolled. Information would be collected on adverse events of subjects enrolled within one year after the implantation of the Bactiseal Catheter from August 07, 2018 to Novemver 30, 2020.

The following information would be collected from subjects' medical records or hospitals' databases (if any):

1. General condition of the subjects
2. Intraoperative condition and catheter implantation
3. Information on the shunt product
4. Adverse events of subjects within one year after the operation and classification of the adverse events
5. Relevant examinations in case of postoperative infection
6. Other adverse event-related information (except anticipated adverse events)

ELIGIBILITY:
Inclusion Criteria:

* The informed consent was exempted by the Ethics Committee of a research center. Either a subject or his/her legal representative signed the informed consent form (ICF) prior to enrollment.
* A subject had an indication suitable to use Bactiseal Catheter.
* A subject received a hydrocephalus shunt at least one year ago.

Exclusion Criteria:

* A subject didn't have an indication suitable to use the product.
* A subject was known to be allergic to a component or ingredient of the product to be implanted, including silicone tubing, rifampicin, and clindamycin.
* According to the comprehensive judgment of an investigator, a subject had an infection of the implant site when the shunt was implanted, such as ventriculitis, meningitis, peritonitis, and local implant skin infection.
* A subject was simultaneously implanted with another shunt system different from Bactiseal Catheter.
* A subject had a contraindication of the shunt operation.
* A subject had uncorrected coagulopathy or any bleeding disorder.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects had an indication suitable to use Bactiseal Catheter and have received a hydrocephalus shunt at least one year ago.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hua Tang, MD, Study Director — Integra Life Sciences
Locations (3):
- China (3):
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Shanghai Children's Medical Center affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in Shanghai Children's Medical Center, School of Medicine, Shanghai Jiao Tong University, Beijing Children Hospital, Capital Medical University, Beijing Hospital. The first subject was enrolled in Sep 1, 2020, and last subject was enrolled in Nov 16, 2020.
Pre-assignment Details: Screened 62 patients, 50 of them were enrolled, including 7 adult patients and 43 minors (subject age below 18). 12 patients were screening failures for not meeting inclusion/exclusion criteria and without post operation follow up.
Groups:
- Bactiseal Catheter Arm: Hydrocephalus subjects implanted with a Bactiseal catheter for one year.
Period: Overall Study
Arm/Group | Bactiseal Catheter Arm
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 50 enrolled subjects were included into PPS
Arm/Group | Bactiseal Catheter Arm
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 43
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: year] | 9.38 [0.11 to 69.96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 50

OUTCOME MEASURES:

1. Primary Outcome: 50 Participants With Non-infection Within One Year
Description: 50 Participants with Non-infection Within One Year
Time Frame: 1 year
Population: 50 participants implanted Bactiseal Catheter for 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bactiseal Catheter Arm
Number analyzed (Participants) | 50
Participants | 1

2. Secondary Outcome: Type and Incidence of Adverse Events of 50 Subjects Within One Year
Description: Type and incidence of adverse events of 50 subjects within one year after catheter implanted
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2043-08

ADVERSE EVENTS:
Time Frame: within 1 year after investigated device implanted
Arm/Group | Bactiseal Catheter Arm
All-Cause Mortality (participants affected / at risk) | 1/50
Serious Adverse Events (participants affected / at risk) | 13/50
Other Adverse Events (participants affected / at risk) | 30/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bactiseal Catheter Arm (N=50)
cerebral hemorrhage (Nervous system disorders) | 2 (2)
subdural hematoma (Nervous system disorders) | 2 (2)
intracranial infection (Nervous system disorders) | 1 (1)
shunt device disorder (Investigations) | 1 (1)
shunt device occlusion (Investigations) | 1 (1)
shunt blockage (Investigations) | 1 (1)
Electrolyte disorders (Metabolism and nutrition disorders) | 1 (1)
Infectious pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1)
Demyelination (Nervous system disorders) | 1 (1)
Infantile spasms (Nervous system disorders) | 1 (1)
Epilepsia (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bactiseal Catheter Arm (N=50)
diarrhea (Gastrointestinal disorders) | 8 (8)
respiratory infection (Respiratory, thoracic and mediastinal disorders) | 6 (6)
fever (Infections and infestations) | 5 (5)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cerebral hemorrhage (Nervous system disorders) | 2 (2)
Subdural hematoma (Nervous system disorders) | 2 (2)
Epilepsia (Nervous system disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT04496414/Prot_SAP_000.pdf